CLINICAL TRIAL: NCT04926103
Title: Screening Donors for a Fecal Microbiota Transplant Program in Ulcerative Colitis: Evaluating Efficacy and Long-term Effects. the FUEL Study
Brief Title: Screening Donors, Fecal Microbiota Transplant Program in Ulcerative Colitis
Acronym: FUEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Paul Moayyedi, Principle Investigator, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUEL001
Record Dates: First submitted 2021-05-12; First posted 2021-06-14 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis Flare
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This is an open label study with all UC patients receiving FMT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label FMT therapy (Experimental): FMT from a related or unrelated healthy donor screened for known communicable disease
  Interventions: Other: Fecal Microbiota transplant (FMT)

INTERVENTIONS:
Other: Fecal Microbiota transplant (FMT) — Patients will come once a week for FMT for 8 weeks. FMT is the administration of the supernatant component of stool and water mixture from a healthy relative or an unrelated donor. The donor's stool and blood is rigorously screened to exclude known communicable diseases. Those that achieve remission with FMT will have the option of continuing FMT once per month for 3 years

SUMMARY:
The investigators intend to screen for new donors, given that there may a donor effect (PubMed ID: 25857665), with some donors not inducing remission in any patient whilst others inducing remission in 20-40% of cases. It is important to give UC patients participating in RCTs stool that has been demonstrated to be effective in some patients. We therefore propose to conduct an open label study in patients with active UC to ensure new donors are effective at inducing remission in some patients. Patients that have FMT will relapse within 18 months (PubMed ID: 25857665) although further FMT therapy induces remission so it is possible that maintenance FMT will result in long term remission, but this needs evaluation. We will therefore follow UC patients that have responded to FMT long term in this open label study.

DETAILED DESCRIPTION:
This is an open label study with all UC patients receiving FMT. Up to 200 patients with active UC will be recruited to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or over
2. Active UC defined as a Mayo score (7) >3
3. A Mayo endoscopic score (7) >0
4. Females of child-bearing potential must be willing and able to use acceptable contraception as per Appendix III. II. b. Toxicity section of the Health Canada Guidance

Exclusion Criteria:

1. Participating in another intervention study for UC
2. Unable to give informed consent
3. Severe comorbid medical illness
4. Severe UC requiring hospitalization.
5. Increase in medical therapy for UC in the last 12 weeks. Continued treatment with 5-ASA, azathioprine, 6-mercaptopurine or anti-TNF therapy (e.g. infliximab) will be permitted if taken at stable dose for ≥12 weeks prior to randomization. Relapse on a stable dose (same dose for at least 2 weeks) or a tapering dose of steroids will also be permitted provided the dose of steroid is not increased again. Stable intake of probiotic therapy also permitted.
6. Antibiotic therapy in the last 30 days.
7. Pregnant women.
8. Patients with clinically significant hepatic dysfunction at the time of screening: ALT > 5 times the upper normal range.
9. Patients with clinically significant renal dysfunction at the time of screening: serum creatinine > 300 µmol/L
10. Any condition, in the opinion of the investigator, that the treatment may pose a health risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of FMT donors at inducing UC remission | 9 weeks
  Suitability of FMT donors at inducing remission in active UC (remission defined as a Mayo score (7) < 3 with an endoscopic Mayo score = 0 at the end of 8 weeks of FMT).
Efficacy of FMT at maintaining remission in UC | 3 years
  Maintenance of remission of UC after three years in those who achieve initial remission with FMT. This is defined as no relapse over three years that requires any medical therapy other than more intense FMT therapy

SECONDARY OUTCOMES:
Efficacy of FMT at in inducing histological remission in active UC | 9 weeks
  Histological remission with no active inflammation on rectal and sigmoid biopsies
Efficacy of FMT at relieving PRO2 symptoms | 9 weeks
  A score of zero on the first two questions of the Mayo Score
Efficacy of FMT at improving Quality of life | 9 weeks and 3 years
  Improvement in quality of life from baseline measured by EQ5D
Adverse effects of FMT | 3 years
  Adverse effects associated with FMT therapy
Stool microbiota predicting FMT success | 9 weeks
  Comparison of stool microbiota evaluated by 16s RNA and metagenomics in those achieving remission with FMT versus those that are not successful
Mucosal microbiota predicting FMT success | 9 weeks
  Comparison of mucosal microbiota evaluated by 16s RNA and metagenomics in those achieving remission with FMT versus those that are not successful

CONTACTS AND LOCATIONS:
Overall Officials: Paul Moayyedi, MD, Principal Investigator — HHSC/McMaster
Locations (1):
- Hamilton Health Sciences / McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Approach investigator to ask for anonymized dataset
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after study completion - estimated 7 years
Access Criteria: Any researcher evaluating the efficacy of FMT in ulcerative colitis

REFERENCES:
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665